CLINICAL TRIAL: NCT01682031
Title: Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase II Trial of Selenomethionine as a Modulator of Efficacy and Toxicity of Chemoradiation in Locally-Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Selenomethionine in Reducing Mucositis in Patients With Locally Advanced Head and Neck Cancer Who Are Receiving Cisplatin and Radiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: I 107807; NCI-2009-01503 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT00935038 (obsolete NCT alias)
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Chemotherapeutic Agent Toxicity; Mucositis; Radiation Toxicity; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Xerostomia
MeSH Terms: conditions — Mucositis; Radiation Injuries; Squamous Cell Carcinoma of Head and Neck; Xerostomia | interventions — Selenomethionine; Cisplatin; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (placebo, cisplatin, and radiotherapy) (Placebo Comparator): Patients receive placebo PO twice daily in week 1 and then once daily in weeks 2-11. Patients also receive cisplatin IV over 3 hours once in weeks 2, 5, and 8 and undergo radiotherapy 5 days a week in weeks 2-8.
  Interventions: Other: placebo; Drug: cisplatin; Radiation: radiation therapy; Procedure: quality-of-life assessment
- Arm II (selenomethionine, cisplatin, and radiotherapy) (Experimental): Patients receive selenomethionine PO twice daily in week 1 and then once daily in weeks 2-11. Patients also receive cisplatin and undergo radiotherapy as in arm I.
  Interventions: Dietary Supplement: selenomethionine; Drug: cisplatin; Radiation: radiation therapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Dietary Supplement: selenomethionine — Given PO
  Arms: Arm II (selenomethionine, cisplatin, and radiotherapy)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm I (placebo, cisplatin, and radiotherapy)
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized phase II trial is studying how well selenomethionine (SLM) works in reducing mucositis in patients with locally advanced head and neck cancer who are receiving cisplatin and radiation therapy. SLM may help prevent or reduce mucositis, or mouth sores, in patients receiving chemotherapy and radiation therapy. It is not yet known whether SLM is more effective than a placebo in reducing mucositis

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether SLM reduces the incidence of grade 3 or 4 mucositis in head and neck squamous cell carcinoma (HNSCC) patients treated with concurrent chemoradiation (CRT) over 7 weeks.

SECONDARY OBJECTIVES:

I. To assess the impact of SLM on tumor complete response rate, relapse-free survival, overall survival and quality of life.

II. To assess whether SLM reduces the incidence and severity of treatment-related toxicities including xerostomia, renal impairment and myelosuppression.

III. To assess whether SLM improves chemoradiation dose delivery. IV. To determine safety of SLM at this dose. V. In New Zealand (NZ) patients only, to assess the impact of SLM on plasma free cisplatin and plasma selenium pharmacokinetics (PK) and on pharmacodynamic (PD) markers of biological activity of selenium.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive placebo orally (PO) twice daily in week 1 and then once daily in weeks 2-11. Patients also receive cisplatin intravenously (IV) over 3 hours once in weeks 2, 5, and 8 and undergo radiotherapy 5 days a week in weeks 2-8.

ARM II: Patients receive selenomethionine PO twice daily in week 1 and then once daily in weeks 2-11. Patients also receive cisplatin and undergo radiotherapy as in arm I.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven locally-advanced HNSCC, including those with cancers of the oral cavity, oropharynx, hypopharynx, larynx, nasopharynx or paranasal sinuses
* Stage III, IVa or IVb disease
* No prior definitive surgery for present diagnosis
* Appropriate candidate for concurrent cisplatin and radiation as definitive treatment; patients who receive induction chemotherapy as part of a definitive treatment program that will include concurrent CRT are eligible for this study
* Hemoglobin >= 10 g/dL (100 g/l)
* Absolute neutrophil count >= 2,000 cells/mm^3 (2 x 10^9/l)
* Platelets >= 100,000 cells/mm^3 (100 x 10^9/l)
* Serum creatinine =< 1.5 mg/dL (133 umol/l) or calculated creatinine clearance >= 50 ml/min using the Cockcroft-Gault formula
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Able to give written informed consent
* Be willing and able to comply with study procedures

Exclusion Criteria:

* Non-regional metastatic disease (stage IVc)
* Previous malignancy within the last 5 years except for adequately treated basal or squamous cell carcinoma of the skin or cervical intra-epithelial neoplasia
* Prior chemotherapy or radiotherapy for HNSCC, or any prior radiotherapy that would compromise delivery of a radical dose to the HNSCC
* Known to be positive for hepatitis C or human immunodeficiency virus (HIV)
* Unable to tolerate oral medication (unless a feeding tube is in place)
* History of hypersensitivity to platinum drugs
* Symptomatic peripheral neuropathy >= National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) grade II
* Pregnant, lactating or unwilling to use adequate contraception
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Planned use of amifostine for prophylaxis against radiation-induced xerostomia
* Patients taking selenium supplements in excess of 100 ug/day
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Evidence of any other significant medical disorder or laboratory finding that in the opinion of the Investigator compromises the subject's safety during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- Roswell Park Cancer Institute, Buffalo, New York, United States
- Waikato Hospital, Hamilton, New Zealand

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Started | 8 | 10
Completed | 7 | 5
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — MRI results indicate increased nodul | 0 | 1
Not completed — Patient could not swallow tablets | 1 | 0
Not completed — Patient stopped selenium on his own | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy) | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (6.6) | 57.4 (8.2) | 57.1 (7.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Incidence of >= Grade 3 Mucositis
Description: Will be compared as difference in proportions with 95% confidence intervals.
Time Frame: Up to 5 years
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Tumor Complete Response Rate
Description: Will be compared as difference in proportions with 95% confidence intervals. Disease will be measured according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Up to 5 years post-treatment
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Relapse-free Survival (RFS)
Description: Assessed by Kaplan-Meier RFS curves and the proportion with an event at 1 year for RFS will be compared simultaneously to obtain more global sensitivity to differences in time-to-event.
Time Frame: At 1 year
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method. Log-rank tests will be used for the comparison of survival distributions among study groups. Continuous endpoints will be summarized using means, standard deviations and percentiles.
Time Frame: Up to 5 years post-treatment
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life
Time Frame: Up to 1 year post-treatment
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Grade 3 or 4 Treatment-related Toxicities, Including Xerostomia
Description: Will be compared as difference in proportions with 95% confidence intervals.
Time Frame: Up to 5 years post-treatment
Population: All treated and eligible patients
Measure: Number; unit: number of xerostomia events
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 8 | 10
number of xerostomia events | 1 | 0

7. Secondary Outcome: CRT Dose Delivery
Description: This characteristic will be included in Cox models.
Time Frame: Up to 8 weeks
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Plasma Cisplatin and Selenium PK and PD Markers (NZ Only)
Description: Descriptive statistics will be used to describe the mean plasma cisplatin and selenium at each time point. Repeated measures analysis of variance will be used to evaluate the changes in plasma cisplatin and selenium over time. Analysis of pharmacodynamic markers will be conducted using statistical methods appropriate for within-patient sequential analyses, such as repeated measures analysis of variance.
Time Frame: Up to 3 months post-treatment
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Placebo, Cisplatin, and Radiotherapy) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy)
Serious Adverse Events (participants affected / at risk) | 4/8 | 2/10
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Placebo, Cisplatin, and Radiotherapy) (N=8) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy) (N=10)
Leukopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Mucosal inflammation (General disorders) | 1 (3) | 1 (3)
Pyrexia (General disorders) | 1 (3) | 0 (0)
Blood creatine increased (Investigations) | 1 (3) | 0 (0)
Blood sodium abnormal (Investigations) | 1 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 1 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Placebo, Cisplatin, and Radiotherapy) (N=8) | Arm II (Selenomethionine, Cisplatin, and Radiotherapy) (N=10)
Leukopenia (Blood and lymphatic system disorders) | 1 (3) | 2 (9)
Lymphopenia (Blood and lymphatic system disorders) | 2 (18) | 3 (27)
White blood cell disorder (Blood and lymphatic system disorders) | 1 (3) | 1 (3)
Angina pectoris (Cardiac disorders) | 1 (3) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (3) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 2 (6) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (3) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (3) | 3 (12)
Diplopia (Eye disorders) | 0 (0) | 1 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (24) | 6 (30)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 3 (21)
Dry mouth (Gastrointestinal disorders) | 5 (15) | 5 (15)
Dysphagia (Gastrointestinal disorders) | 5 (21) | 5 (15)
Glossodynia (Gastrointestinal disorders) | 1 (3) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (3)
Mouth ulceration (Gastrointestinal disorders) | 1 (3) | 1 (3)
Nausea (Gastrointestinal disorders) | 5 (24) | 8 (27)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (6)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (3) | 1 (3)
Oral pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (6)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (9) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (3) | 2 (6)
Vomiting (Gastrointestinal disorders) | 3 (9) | 2 (6)
Asthenia (General disorders) | 0 (0) | 1 (3)
Fatigue (General disorders) | 5 (21) | 6 (39)
Fibrosis (General disorders) | 1 (3) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 2 (6)
Mucosal inflammation (General disorders) | 4 (24) | 6 (30)
Oedema peripheral (General disorders) | 1 (3) | 1 (3)
Pain (General disorders) | 1 (3) | 1 (3)
Pyrexia (General disorders) | 2 (6) | 2 (6)
Secretion discharge (General disorders) | 1 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (3)
Oral candidiasis (Infections and infestations) | 1 (3) | 1 (3)
Perianal abscess (Infections and infestations) | 0 (0) | 1 (3)
Radiation skin injury (Injury, poisoning and procedural complications) | 4 (15) | 3 (9)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3)
Blood bilirubin abnormal (Investigations) | 0 (0) | 1 (6)
Blood creatine increased (Investigations) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 1 (6) | 0 (0)
Blood sodium abnormal (Investigations) | 1 (3) | 0 (0)
Haemoglobin (Investigations) | 1 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (9) | 4 (27)
Neutrophil count decreased (Investigations) | 2 (6) | 1 (3)
Platelet count decreased (Investigations) | 1 (3) | 2 (9)
Weight decreased (Investigations) | 2 (6) | 2 (9)
White blood cell count decreased (Investigations) | 0 (0) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (18) | 3 (12)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 3 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (15) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (6) | 1 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (21) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (6) | 4 (18)
Oral intake reduced (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (6)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (3)
Dysgeusia (Nervous system disorders) | 4 (12) | 6 (21)
Facial paresis (Nervous system disorders) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (12) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (6) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 2 (9)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 2 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (3)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (18)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (18) | 6 (24)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (6)
Erythema (Skin and subcutaneous tissue disorders) | 4 (18) | 7 (30)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (6) | 0 (0)
Thrombosis (Vascular disorders) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes